CLINICAL TRIAL: NCT06106867
Title: The Effect of External Pressure Applı̇ed to the Palm on Labor Paı̇n and Childbirth Experı̇ence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Emine Nur Çalımlı Celep, Principal Investigator, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IUC-ENC
Record Dates: First submitted 2023-10-04; First posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Labor Pain
Keywords: external pressure; labor pain; childbirth experience; non-pharmacological method; midwifery care
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Information about applying external pressure to the palm was provided to the pregnant women in the experimental group. The researcher practically explained how, when and for how long to apply external pressure to the palm. The researcher introduced the comb to be used in the application of external pressure to the palm, and the application stage of the study was started.
  Interventions: Procedure: External pressure to the palm
- Control Group (No Intervention): Routine midwifery care and services applied to all pregnant women in the hospital were provided to the participants in the control group.

INTERVENTIONS:
Procedure: External pressure to the palm — During the 5-6 cm, 7-8 cm, and 9-10 cm cervical dilatation stages of the labor process, palm external pressure was applied to the pregnant women in the experimental group.
  Arms: Experimental Group

SUMMARY:
The study was carried out to evaluate the effect of external pressure applied to the palm on labor pain and childbirth experience.The sample of the randomized controlled study consisted of 60 nulliparous (30 in the experimental group and 30 in the control group) pregnant women who presented to Zeynep Kamil Gynecology and Pediatrics Training and Research Hospital between April and June 2020 to give birth and met the research conditions. The Descriptive Information Form, Follow-Up Form Related to Labor Action, Childbirth Experience Questionnaire (CEQ), and Visual Analogue Scale (VAS) were used in data collection. During the 5-6 cm, 7-8 cm, and 9-10 cm cervical dilatation stages of the labor process, palm external pressure was applied to the pregnant women in the experimental group, while standard midwifery care was provided to the pregnant women in the control group. The VAS was applied to both groups at admission to the hospital, before and after the 5-6 cm, 7-8 cm, and 9-10 cm cervical dilatation stages, and also at the 30th minute postpartum. Data were analyzed Statistical Package for Social Sciences 24.0 program using number, percentage, mean, standard deviation, the Kolmogorov-Smirnov test, Levene's test and independent samples t-test, one-way ANOVA test, analysis of variance, and chi-square test. In all analyses, p<0.05 values will be considered statistically significant.

DETAILED DESCRIPTION:
Labor pain adversely affects pregnant women's perception of the labor process and childbirth. When not taken under control, it causes pregnant women to have negative experiences about the labor process and consequently leads to a decrease in their satisfaction with childbirth. For this reason the study was carried out to evaluate the effect of external pressure applied to the palm on labor pain and childbirth experience. Hypotheses of the research; H 1 : External pressure applied to the palm during labor reduces the level of labor pain. H 1 : External pressure applied to the palm during labor increases the positive birth experience.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 18-35 years
* Being a nulliparous pregnant woman
* Being pregnant at term (between the 37th and 42nd weeks of gestation)
* Expecting the vaginal delivery
* Being in singleton and vertex presentation
* The weight of the fetus between 2500-4000 g
* Having had an uncomplicated pregnancy process for the pregnant woman and the fetus
* Being in the latent phase (cervical dilatation below 4 cm)

Exclusion Criteria:

* Having high-risk pregnancy
* Having any disease and disability related to the hand and palm
* Having any health problem preventing communication
* Being a pregnant woman in need of analgesics
* Pregnant women to whom non-pharmacological methods were applied to relieve pain
* Undergoing cesarean section due to possible indication

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 60 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) Level of labor pain will be measured with VAS. | 30 minutes
  (min:0, max:10)
The Childbirth Experience Questionnaire (CEQ) | At the 30th minute postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Emine Nur Çalımlı Celep, Principal Investigator — Researcher Assistant
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abdul-Sattar Khudhur Ali S, Mirkhan Ahmed H. Effect of Change in Position and Back Massage on Pain Perception during First Stage of Labor. Pain Manag Nurs. 2018 Jun;19(3):288-294. doi: 10.1016/j.pmn.2018.01.006. Epub 2018 Apr 19. PMID 29680213
- [Background] ACOG Committee Opinion No. 766: Approaches to Limit Intervention During Labor and Birth. Obstet Gynecol. 2019 Feb;133(2):e164-e173. doi: 10.1097/AOG.0000000000003074. PMID 30575638
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Bodian CA, Freedman G, Hossain S, Eisenkraft JB, Beilin Y. The visual analog scale for pain: clinical significance in postoperative patients. Anesthesiology. 2001 Dec;95(6):1356-61. doi: 10.1097/00000542-200112000-00013. PMID 11748392
- [Background] Chaillet N, Belaid L, Crochetiere C, Roy L, Gagne GP, Moutquin JM, Rossignol M, Dugas M, Wassef M, Bonapace J. Nonpharmacologic approaches for pain management during labor compared with usual care: a meta-analysis. Birth. 2014 Jun;41(2):122-37. doi: 10.1111/birt.12103. Epub 2014 Apr 25. PMID 24761801
- [Background] Dencker A, Taft C, Bergqvist L, Lilja H, Berg M. Childbirth experience questionnaire (CEQ): development and evaluation of a multidimensional instrument. BMC Pregnancy Childbirth. 2010 Dec 10;10:81. doi: 10.1186/1471-2393-10-81. PMID 21143961
- [Background] Jones L, Othman M, Dowswell T, Alfirevic Z, Gates S, Newburn M, Jordan S, Lavender T, Neilson JP. Pain management for women in labour: an overview of systematic reviews. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD009234. doi: 10.1002/14651858.CD009234.pub2. PMID 22419342
- [Background] Lang AJ, Sorrell JT, Rodgers CS, Lebeck MM. Anxiety sensitivity as a predictor of labor pain. Eur J Pain. 2006 Apr;10(3):263-70. doi: 10.1016/j.ejpain.2005.05.001. Epub 2005 Jun 28. PMID 15987671
- [Background] Myles PS. The pain visual analog scale: linear or nonlinear? Anesthesiology. 2004 Mar;100(3):744; author reply 745. doi: 10.1097/00000542-200403000-00042. No abstract available. PMID 15108996
- [Background] Smith CA, Levett KM, Collins CT, Jones L. Massage, reflexology and other manual methods for pain management in labour. Cochrane Database Syst Rev. 2012 Feb 15;(2):CD009290. doi: 10.1002/14651858.CD009290.pub2. PMID 22336862
- [Background] Soriano-Vidal FJ, Oliver-Roig A, Cabrero-Garcia J, Congost-Maestre N, Dencker A, Richart-Martinez M. The Spanish version of the Childbirth Experience Questionnaire (CEQ-E): reliability and validity assessment. BMC Pregnancy Childbirth. 2016 Nov 24;16(1):372. doi: 10.1186/s12884-016-1100-z. PMID 27884123
- [Background] WHO recommendations: Intrapartum care for a positive childbirth experience. Geneva: World Health Organization; 2018. Available from http://www.ncbi.nlm.nih.gov/books/NBK513809/ PMID 30070803
- [Result] Hamidzadeh A, Shahpourian F, Orak RJ, Montazeri AS, Khosravi A. Effects of LI4 acupressure on labor pain in the first stage of labor. J Midwifery Womens Health. 2012 Mar-Apr;57(2):133-8. doi: 10.1111/j.1542-2011.2011.00138.x. Epub 2012 Mar 2. PMID 22432484
- [Result] Rosseland LA, Reme SE, Simonsen TB, Thoresen M, Nielsen CS, Gran ME. Are labor pain and birth experience associated with persistent pain and postpartum depression? A prospective cohort study. Scand J Pain. 2020 Jul 28;20(3):591-602. doi: 10.1515/sjpain-2020-0025. PMID 32469334
- [Result] Sehhatie-Shafaie F, Kazemzadeh R, Amani F, Heshmat R. The effect of acupressure on sanyinjiao and hugo points on labor pain in nulliparous women: a randomized clinical trial. J Caring Sci. 2013 Jun 1;2(2):123-9. doi: 10.5681/jcs.2013.015. eCollection 2013 Jun. PMID 25276718
- [Result] Smith CA, Levett KM, Collins CT, Dahlen HG, Ee CC, Suganuma M. Massage, reflexology and other manual methods for pain management in labour. Cochrane Database Syst Rev. 2018 Mar 28;3(3):CD009290. doi: 10.1002/14651858.CD009290.pub3. PMID 29589380